CLINICAL TRIAL: NCT04009525
Title: Hematopoietic Stem Cell Transplantation for Patients With Thalassemia Major: A Multicenter, Prospective Clinical Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: Peking University People's Hospital (Other); Ruijin Hospital (Other); The 923rd Hospital of Joint Logistics Support Force of People's Liberation Army (Other); LiuZhou People's Hospital (Other); The First People's Hospital of Yunnan (Other); Liuzhou Workers' Hospital (Other Government); Xinqiao Hospital of Chongqing (Other); Affiliated Hospital of Youjiang University of Ethnic Medicine (Unknown); Hainan People's Hospital (Other); Maoming People's Hospital (Other); Red Cross Hospital of Yulin City (Other); Guilin Medical College (Other); Wuzhou People's Hospital (Unknown); Guangxi Autonomous Region People's Hospital (Unknown); The 920th Hospital of Joint Logistics Support Force of People's Liberation Army (Unknown)
Responsible Party: Principal Investigator, Yongrong Lai, Director of the Hematology Department, First Affiliated Hospital of Guangxi Medical University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GX-HSCT-MT 2019
Record Dates: First submitted 2019-07-03; First posted 2019-07-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Thalassemia Major
Keywords: thalassemia major; hematopoietic stem cell transplantation
MeSH Terms: conditions — beta-Thalassemia | interventions — Busulfan; Cyclophosphamide; fludarabine; Influenza Vaccines; thymoglobulin; Cyclosporine; Mycophenolic Acid; Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MSD-HSCT (Experimental): matched sibling donors hematopoietic stem cell transplantation
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Thymoglobulin; Drug: cyclosporine A; Drug: Mycophenolate mofetil; Drug: Methotrexate
- URD-HSCT (Experimental): unrelated donor hematopoietic stem cell transplantation
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Thymoglobulin; Drug: Mycophenolate mofetil; Drug: Tacrolimus; Drug: Methotrexate
- haplo-HSCT (Experimental): haplo-identical hematopoietic stem cell transplantation
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Thymoglobulin; Drug: Mycophenolate mofetil; Drug: Tacrolimus; Drug: Methotrexate

INTERVENTIONS:
Drug: Busulfan — Busulfan（4 mg/kg/day,4 days）
  Other Names: Bu
Drug: Cyclophosphamide — Cyclophosphamide（50 mg/kg/day,4 days）
  Other Names: Cy
Drug: Fludarabine — Fludarabine（50 mg/m2/day,3 days）
  Other Names: Flu
Drug: Thymoglobulin — Thymoglobulin（2.5 mg/kg/day,4 days）
  Other Names: ATG
Drug: cyclosporine A — cyclosporine A
  Other Names: CsA
  Arms: MSD-HSCT
Drug: Mycophenolate mofetil — Mycophenolate mofetil（0.25g/day）
  Other Names: MMF
Drug: Tacrolimus — Tacrolimus
  Other Names: FK506
  Arms: URD-HSCT; haplo-HSCT
Drug: Methotrexate — Methotrexate
  Other Names: MTX

SUMMARY:
The only curative therapy for thalassemia major remains the replacement of the defective erythropoiesis by allogeneic hematopoietic stem cell transplantation(allo-HSCT). We conduct a prospective multicenter study to evaluate the efficacy of allo-HSCT in the treatment of thalassemia major.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is one of the established curative option for thalassemia major (TM). Previous study has predicted that more than 90% of TM patients can survive after allo-HSCT with a thalassemia-free survival (TFS) in around 80% of them.The purpose of this study is to evaluate the efficacy of allo-HSCT in the treatment of thalassemia major.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with thalassemia major.
2. Indication of hematopoietic stem cell transplantation.
3. A cardiac ejection fraction of >50%; normal pulmonary function tests and pulmonary examination results; and normal kidney function.

Exclusion Criteria:

1. Aspartate aminotransferase levels > 4-fold the upper limit of the normal range for our institution's lab criteria;
2. Uncontrolled bacterial, viral or fungal infections;
3. Any other restriction for transplantation.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 823 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years
  2-years overall survival
Thalassemia-free survival | 2 years
  2-years thalassemia-free survival

SECONDARY OUTCOMES:
Engraftment | 30 days
  Myeloid engraftment at day +30
Transplant Related Mortality | 2 year
  Transplant-related mortality by 2 year
Cumulative Incidence of acute Graft Versus Host Disease | 100 days
  Acute graft versus host disease at day +100
Cumulative Incidence of chronic Graft Versus Host Disease | 2 years
  Chronic graft versus host disease by 2 years
Cumulative Incidence of Infectious Complications | 2 years
  Cumulative incidence of bacterial, fungal and viral infections by 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yongrong Lai, MD, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China